CLINICAL TRIAL: NCT01951326
Title: A Randomized, Double Blind, Placebo-controlled, Multicenter, Parallel Group Study to Assess the Efficacy and Safety of Fixed-dose Combination RHB-104 in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: Efficacy and Safety of Anti-MAP Therapy in Adult Crohn's Disease
Acronym: MAPUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHB-104-01
Record Dates: First submitted 2013-09-19; First posted 2013-09-26 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-06

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; moderate to severe; remission; MAP; antibiotic
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RHB-104 (Active Comparator): 5 RHB-104 capsules administered orally BID
  Interventions: Drug: RHB-104
- Placebo (Placebo Comparator): 5 placebo capsules administered orally BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RHB-104 — 95 mg clarithromycin, 45 mg rifabutin, and 10 mg clofazimine
  Arms: RHB-104
Drug: Placebo — 5 placebo capsules administered orally BID
  Arms: Placebo

SUMMARY:
The investigators hypothesize that RHB-104 will have greater efficacy than placebo in Crohn's disease.

DETAILED DESCRIPTION:
A Randomized, Double Blind, Placebo-controlled, Multicenter, Parallel Group Study to Assess the Efficacy and Safety of Fixed-dose Combination RHB-104 in Subjects with Moderately to Severely Active Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria

1. Signed fully informed consent provided as per this protocol.
2. Diagnosis of Crohn's Disease confirmed by endoscopy or radiography and/or histology at least 6 months prior to randomization into the study.
3. CD involving the ileum and/or colon
4. Moderately to severely active CD (Crohn's Disease Activity Index (CDAI) score of greater than or equal to 220 and less than or equal to 450) at baseline.
5. Current treatment with at least one of the following therapies:

   A. Oral 5-acetyl salicylic acid (5-ASA) compounds. Dose must be stable for at least 4 weeks before baseline.

   B. Corticosteroid therapy. Dose must be stable for at least 2 weeks before baseline.

   C. Azathioprine or 6-mercaptopurine (6-MP) or methotrexate. Dose must be stable for at least 8 weeks before baseline.

   D. Infliximab or adalimumab. Dose must be stable for at least 14 weeks before baseline.
6. White blood cell count greater than or equal to 3.5 x 109 at screening.
7. Active Crohn's disease, defined by at least one of the following: C-reactive protein greater than Upper Limit of Normal (ULN) at screening, fecal calprotectin greater than Upper Limit of Normal (ULN) at screening, OR radiographic (MRE or CTE) or endoscopic confirmation of the presence of active CD within 5 weeks of screening visit. .
8. Subject agrees to use barrier contraceptive methods (i.e. diaphragm, cervical cap, contraceptive sponge or condom) with spermicidal foam/gel/cream/suppository, IUD/IUS or progestogen injection (Depo-Provera®) throughout the study and for at least 6 weeks after last study drug administration, unless subject is post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation, or has had a vasectomy. In regions where local regulatory contraceptive requirements differ, the ICF will reflect local policies.

Exclusion Criteria

1. Crohn's Disease involvement isolated to the mouth, upper gastrointestinal tract, or anus.
2. History of total colectomy with ileorectal anastomosis or a proctocolectomy.
3. Presence of active fistulizing Crohn's Disease or healed fistula within 2 months prior to screening.
4. Subject has postoperative stoma, ostomy, or ileoanal pouch.
5. Subject has short bowel syndrome.
6. Subject is scheduled for surgical bowel resection.
7. Subject has known symptomatic obstructive strictures or bowel perforation in the 6 months prior to screening.
8. Change in dose or discontinuation of oral 5-acetyl salicylic acid (5-ASA) compounds less than 4 weeks prior to baseline.
9. Change in dose or discontinuation of corticosteroids less than 2 weeks prior to baseline.
10. Change in dose or discontinuation of azathioprine, 6-mercaptopurine (6-MP) or methotrexate less than 8 weeks prior to baseline.
11. Change in dose or discontinuation of infliximab or adalimumab less than 14 weeks prior to baseline.
12. Treatment with vedolizumab less than 120 days prior to baseline or biological therapies (apart from infliximab or adalimumab) less than 60 days prior to baseline.
13. Previous treatment with rifabutin and/or clofazimine.
14. Oral or parenteral antibiotics in the 4 weeks prior to baseline (topical antibiotics are permitted).
15. Treatment with probiotics (excluding yogurt and yogurt-derived products) in the 4 weeks prior to baseline.
16. Females who have a positive pregnancy test or are lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2013-09; Primary Completion 2018-05 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira N Kalfus, MD, Study Director — RedHill Biopharma; David Y. Graham, MD, Principal Investigator — Department of Medicine/Gastroenterology, Baylor College of Medicine, Houston
Locations (103):
- United States (43):
  - Del Sol Research Management, 850 N Knob Road, Tucson, Arizona
  - Associated Gastroenterology Medical Group, 1211 W. La Palmak Ave, Suite 303, Anaheim, California
  - Medvin Clinical Research, 15627 Imperial Highway,, La Mirada, California
  - Digestive Care Associates, Inc., 1000 Laurel St., San Carlos, California
  - Ventura Clinical Trials, 1835 Knoll Drive, Ventura, California
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Innovative Medical Research of South Florida, 2999 NE 191 St., Suite 330, Aventura, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Sunrise Medical Research, Inc. 4700 N. State Road Building A, Suite 111, Lauderdale Lakes, Florida
  - Gastroenterology Group of Naples, 1064 Goodlette Road, Naples, Florida
  - Advanced Research Institute Inc., 7114 Congress Street, New Port Richey, Florida
  - Endoscopic Research, Inc., 1817 North Mills Avenue, Orlando, Florida
  - Advanced Medical Research Center, 1690 Dunlawton Ave., Suite 110, Port Orange, Florida
  - Atlanta Center for Gastroenterology 2665 North Decatur Road Suite 550, Decatur, Georgia
  - Gastrointestinal Specialists of Georgia PC, 711 Canton Rd. Suite 300, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - The Carle Foundation, 611 West Park Street, Urbana, Illinois
  - Cotton-O'Neil Clinical Research Center, 720 SW Lane St., Topeka, Kansas
  - Investigative Clinical Research, 612 Ridgely Avenue, Suite 401,, Annapolis, Maryland
  - Chevy Chase Clinical Research, 5550 Friendship Blvd., Chevy Chase, Maryland
  - Commonwealth Clinical Studies, 189 Quincy St., Brockton, Massachusetts
  - Center For Digestive Health, Troy, Michigan
  - West Michigan Clinical Research Center, 2093 Health Dr. SW, Suite 201, Wyoming, Michigan
  - Ehrhardt Clinical Research, LLC, 108 Congress Street, Belton, Missouri
  - AGA Clinical Research Associates, Inc., 3205 Fire Road, Egg Harbor, New Jersey
  - Holy Name Medical Center, 718 Teaneck Road, Teaneck, New Jersey
  - North Shore Long Island Jewish Medical Group, 600 Northern Boulevard, Suite 111, Great Neck, New York
  - NYU Langone Long Island , 1000 Northern Boulevard, Suite 160, Great Neck, New York
  - Manhattan Medical Research Practice PLLC, 215 Lexington Avenue, 21st Floor, New York, New York
  - Montefiore Medical Center, 111 East 210th Street, The Bronx, New York
  - University of North Carolina Center for inflammatory Bowel Diseases, CB 7080, 130 Mason Farm Road, 4151 Bioinformatics Bldg., Chapel Hill, North Carolina
  - Ohio GI and Liver Institute, 2925 Vernon Place 100, Cincinnati, Ohio
  - Ohio GI and Liver Institute, Cincinnati, Ohio
  - ClinSearch, 6035 Shallowford Road, Suite 109, Chattanooga, Tennessee
  - Brooke Army Medical Center, 3551 Roger Brooke Drive, Fort Sam Houston, Texas
  - Baylor College of Medicine, 7200 Cambridge Street Suite 180.184, 10th Floor, Houston, Texas
  - University of Texas Health Sciences Center at Houston, 6431 Fannin Street, Medical School Bldg 4-234, Houston, Texas
  - Spring Gastroenterology Associates, 8901 FM 1960 West, Humble, Texas
  - DHAT Research Institute / Digestive Health Associates of Texas 3600 Shire Blvd, Suite 106, Richardson, Texas
  - Digestive Disease Center, 621 Camden Street, Suite 202, San Antonio, Texas
  - Tyler Research Institute, 1720 S. Beckham, Tyler, Texas
  - Gasteroenterology Associates of Northern Virgina, 3028 Javier Road, Fairfax, Virginia
  - McGuire DVAMC, 1201 Broad Rock Boulevard, Richmond, Virginia
- Australia (9):
  - Bankstown Hospital, Level 3, Department of Gastroenterology, Eldridge Road, Bankstown, New South Wales
  - Department of Gastroenterology and Hepatology, Concord Hospital, Hospital Road, Concord, New South Wales
  - Nepean Hospital, Derby Street, Kingswood, New South Wales
  - Department of Gastroenterology, Level 1, Clinic 123, New Clinical Building, Liverpool Hospital, Elizabeth St., Liverpool, New South Wales
  - Department of Gastroenterology and Hepatology, Level 9, Ned Hanlon Building, Royal Brisbane and Women's Hospital Corner Butterfield Street and Bowen Bridge Street, Herston, Queensland
  - Mater Hospital Brisbane, Department of Gastroenterology, Raymond Terrace, South Brisbane, Queensland
  - Ballarat Health Services, Drummond St North, Ballarat, Victoria
  - Department of Gastroenterology, Eastern Health, ECRU, Level 2, 5 Arnold Street, Box Hill, Victoria
  - Department of Gastroenterology and Hepatology, Cabrini Medical Centre, 183 Wattletree Road, Malvern, Victoria
- Bulgaria (5):
  - MHAT "Sv. Karidad" EAD, Department of Internal Medicine / Gastroenterology, endocrinology and metabolic disorders, 23А, Nikola Vaptsarov Blvd, Plovdiv
  - MHAT "Hadzhi Dimitar" OOD, Department of Internal Medicine / Gastroenterology and Endocrinology, 5, Dimitar Pehlivanov str., Sliven
  - UMHAT "Sv. Ivan Rilski" EAD; Clinic of Gastroenterology, 15, Akad. Ivan Geshov Blvd.,, Sofia
  - ACIBADEM CITY CLINIC UNIVERSITY HOSPITAL EOOD, Oncology Center, Clinic of Gastroenterology, 66 A, Tsarigradsko shosse Blvd, Sofia
  - DCC "Mladost-M Varna" OOD, office 528 V, 15, Republika Blvd., Varna
- Canada (4):
  - Discovery Clinical Services Ltd. 601 A Discovery St., Victoria, British Columbia
  - Mount Sinai Hospital, 600 University Avenue, Suite 445, Toronto, Ontario
  - Montreal General Hospital Digestive Lab Research Institute McGill University Health Center, 1650 Cedar Avenue C10.145, Montreal, Quebec
  - University of Saskatchewan Royal University Hospital, 103 Hospital Drive IBD Clinical Trials Unit Rm 2658, Saskatoon, Saskatchewan
- Czechia (7):
  - Nemocnice Horovice, NH Hospital, a.s., Chirurgicke oddeleni, K Nemocnici 1106, Hořovice
  - Gastroenterologie s.r.o., Manesova 646,, Hradec Králové
  - HEPATO-GASTROENTEROLOGIE HK, s.r.o., Trida Edvarda Benese 1549/34, Hradec Králové
  - EGK s.r.o., Sanatorium sv. Anny, Gastroenterologicke oddeleni, Lucni 7a/2776,, Prague
  - IBD centrum / ISCARE IVF a.s., Jankovcova 1569/2c, Prague
  - ARTROSCAN, s.r.o., Gastroenterologicka ambulance, 5114 Trebovicka, Ostrava, Třebovice
  - Krajska zdravotni, a.s., Masarykova nemocnice o.z. Gastroenterologie, Socialni pece 3316/12A, Ústí nad Labem
- Israel (10):
  - Assaf HaRofeh Medical Center, Gastroenterology Department, Harofeh Medical Center, Be’er Ya‘aqov
  - Bnaizion Medical Center, Golomb 47, Haifa
  - The E. Wolfson Medical Center, 62 Halohamim Str., Holon
  - Shaare Zedek Medical Center, Beith Street, Jerusalem
  - Ein Karem Medical Center, Kiryat Hadassah, Jerusalem
  - Meir, 59 Tchemacovsky St, Kfar Saba
  - Galilee Medical Center, P.O.B. 21, Nahariya
  - Holy Family Hospital, Namsawi St. POB 8, Nazareth
  - RMC Beilinson Hospital, 39 Jabotinsky Street, Petah Tikva
  - Sourasky Medical Center, 6 Weizman Street, Tel Aviv
- New Zealand (5):
  - Shakespeare Specialist Group, North Shore, Suite 3, 181 Shakespeare Road, Milford Takapuna, Auckland
  - Christchurch Hospital, Christchurch
  - Gastroenterology Unit, Southern District Health Board, 201 Great King Street,, Dunedin
  - Department of Gastroenterology,Waikato Hospital, Hamilton
  - Clinical Trials Unit, Tauranga Hospital,, Tauranga
- Poland (10):
  - NZOZ Specjalistyczne Centrum Gastrologii GASTROMED Wiejska 81, Bialystok
  - SP ZOZ MSWiA w Gdańsku, Oddział Gastroenterologiczny, ul. Kartuska 4/6, Gdansk
  - UNICARDIA Specjalistyczne Centrum Leczenia Chorob Serca i Naczyn & UNIMEDICA Specjalistyczne Centrum Medyczne Sp. z o.o. Kluczborska 15, Krakow
  - Centrum Medyczne Szpital Sw. Rodziny Sp. z o.o. Wigury 19, Lodz
  - Wojewodzki Szpital Kliniczny w Olsztynie Oddzial Gastroenterologiczny Żołnierska 18, Olsztyn
  - ENDOSKOPIA sp. z o.o. B. Chrobrego 6/8, Sopot
  - EuroMedis sp. z.o.o., ul. Powstanców Wielkopolskich 33a, Szczecin
  - "GASTROMED" Kopon, Zmudzinski i wspolnicy sp. j., Specjalistyczne Centrum Gastroskopii i Endoskopii, Specjalistyczne Gabinety Lekarskie Grudziadzka 11, Torun
  - Centralny Szpital Kliniczny MSW w Warszawie Klinika Chorob Wewnetrznych i Gastroenterologii Woloska 137, Warsaw
  - ARS MEDICA s.c. Rybak Maria, Rybak Zbigniew, Powstancow Slaskich 56A/2, Wroclaw
- Serbia (5):
  - : Clinic for Gastroenterology and Hepatology, Clinical Center of Serbia Koste Todorovica 2, Belgrade
  - Clinical Department of Gastroenterology and Hepatology, Clinic for Internal Diseases, Clinical Hospital Center Zvezdara Dimitrija Tucovica 161, Belgrade
  - Department of Gastroenterology and Hepatology, Clinical Hospital Center Zemun Vukova 9, Belgrade
  - : Center for Gastroenterohepatology, Clinic for Internal Medicine, Clinical Center of Kragujevac Zmaj Jovina 30, Kragujevac
  - : Clinic of Gastroenterology and Hepatology, Clinical Center of Vojvodina Hajduk Veljkova 1, Novi Sad
- Slovakia (5):
  - Univerzitna nemocnica Bratislava - Nemocnica Ružinov, V. Interná klinika LFUK a UNB, Gastroenterologické a hepatologické oddelenie, Ruzinovska 6, Bratislava
  - Univerzitná nemocnica Bratislava - Nemocnica sv. Cyrila a Metoda Gastroenterologická klinika SZU a UNB Antolská 11, Bratislava
  - Breznianske centrum gastroenterologie, s.r.o. Banisko 1, Brezno
  - PIGEAS s.r.Prieložtek 1, o.,, Martin
  - KM Management spol. s.r.o., Gastroenterologické a hepatologické centrum Nitra, Špitálska 13, Nitra

REFERENCES:
- [Derived] Graham DY, Naser SA, Borody T, Hebzda Z, Sarles H, Levenson S, Hardi R, Arlukowicz T, Svorcan P, Fathi R, Bibliowicz A, Anderson P, McLean P, Fehrmann C, Harris MS, Zhao S, Kalfus IN. Randomized, Double-Blind, Placebo-Controlled Study of Anti-Mycobacterial Therapy (RHB-104) in Active Crohn's Disease. Antibiotics (Basel). 2024 Jul 25;13(8):694. doi: 10.3390/antibiotics13080694. PMID 39199994
- See also: Related Info — http://www.redhillbio.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RHB-104 | Placebo
Started | 166 | 165
Completed | 87 | 87
Not Completed | 79 | 78

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RHB-104 | Placebo | Total
Number analyzed (Participants) | 166 | 165 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (12.51) | 39.3 (12.56) | 39.1 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 67 | 142
  Male | 91 | 98 | 189
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 12 | 20
  White | 156 | 150 | 306
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Europe | 47 | 50 | 97
  Israel | 18 | 20 | 38
  Southeast Asia | 9 | 12 | 21
  North America | 92 | 83 | 175
Baseline Crohn's Disease Activity Index (CDAI) score [Mean (Standard Deviation); unit: units on a scale] — Generally, CDAI scores can range from 0 to ~600. (in this protocol up to 450)
  CDAI scores of 150-219 describe mildly active disease, while scores of 220-450 describe moderately active disease and scores above 450 describe severe disease.
  units on a scale | 297.77 (57.023) | 293.44 (53.184) | 295.61 (55.102)
Anti-TNF Use at Baseline [Count of Participants; unit: Participants] | 37 | 41 | 78

OUTCOME MEASURES:

1. Primary Outcome: Remission at Week 26
Description: Reduction of the total Crohn's Disease Activity Index (CDAI) score to less than 150. Lower CDAI scores indicate a better outcome.
Time Frame: Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 166 | 165
Participants | 61 | 37
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0048, Cochran-Mantel-Haenszel; Stratified according to anti-TNF agent use (Y/N)

2. Secondary Outcome: Response at Week 26
Description: Reduction of Crohn's Disease Activity Index (CDAI) score by a minimum of 100 points. Lower CDAI scores indicate a better outcome.
Time Frame: Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 166 | 165
Participants | 73 | 50
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0116, Cochran-Mantel-Haenszel; Stratified according to anti-TNF agent use (Y/N)

3. Secondary Outcome: Remission at Week 52
Description: as for outcome 1
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 166 | 165
Participants | 47 | 32
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0616, Cochran-Mantel-Haenszel; Stratified according to anti-TNF agent use (Y/N)

4. Secondary Outcome: Durable Remission Week 26 Through Week 52
Description: When a subject is in remission with a maximum CDAI score of 149 at every visit from Week 26 through and including Week 52
Time Frame: Week 26 through week 52
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 166 | 165
Participants | 33 | 21
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0851, Cochran-Mantel-Haenszel; Stratified according to anti-TNF agent use (Y/N)

5. Secondary Outcome: Remission at Week 16
Description: as for outcome 1
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 166 | 165
Participants | 70 | 48
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0147, Cochran-Mantel-Haenszel; Stratified according to anti-TNF agent use (Y/N)

6. Secondary Outcome: Steroid Free Remission at Week 52
Description: Subjects who are maintained off steroids for a minimum of 3 weeks
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 57 | 55
Participants | 11 | 5
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.1510, Cochran-Mantel-Haenszel; Stratified according to anti-TNF agent use (Y/N)

7. Other Pre Specified Outcome: Duration of Remission
Description: Number of weeks that a subject is in a state of remission. Subjects who experienced remission and continued to be in remission at the time of their last CDAI assessment are censored at the date of their last CDAI assessment.
Time Frame: Baseline through week 52
Population: Reached duration of remission (dropped out of remission during the study), n (%): RHB-104 54 (53.5); Placebo: 49 (62.8). Censored (remain in remission during the study), n (%): RHB-104: 47 (46.5); Placebo 29 (37.2)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 101 | 78
weeks | 27.1 [16.14 to 46.86] | 16.7 [10.14 to 30.00]
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.2402, Log Rank

8. Other Pre Specified Outcome: Duration of Response
Description: Number of weeks a subject is in a state of response. Subjects who experienced response and continued to be in response at the time of their last CDAI assessment are censored at the date of their last CDAI assessment.
Time Frame: Baseline through week 52
Population: Reached duration of response (dropped out of response during the study), n (%) RHB-104: 52 (45.2); Placebo: 55 (59.8). Censored (remain in response during the study), n (%): RHB-104: 63 (54.8); Placebo: 37 (40.2)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 115 | 92
weeks | 40.1 [22.14 to 52.29] | 22.1 [12.14 to 32]
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0460, Log Rank

9. Other Pre Specified Outcome: Time to Remission
Description: [Date of first observed remission (CDAI score < 150) - Date of first dose or date of randomization if not dosed + 1] / 7 Days. Subjects who never experienced remission during the study are censored at the date of their last CDAI assessment.
Time Frame: Baseline through week 52
Population: Number of subjects achieved remission, n (%) RHB-104: 101 (60.8); Placebo 78 (47.3). Censored, n (%): RHB-104: 65 (39.2); Placebo 87 (52.7)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 166 | 165
weeks | 12.1 [8.43 to 12.71] | 19.9 [13.00 to 52.43]
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0031, Log Rank

10. Other Pre Specified Outcome: Time to Response
Description: [Date of first observed response (a reduction from baseline of ≥ 100 in CDAI score) - Date of first dose or date of randomization if not dosed + 1] / 7 Days. Subjects who never experienced response during the study are censored at the date of their last CDAI assessment.
Time Frame: Baseline through week 52
Population: Number of subjects achieved response, n (%): RHB-104: 115 (69.3); Placebo: 92 (55.8); Censored, n (%): RHB-104: 51 (30.7); Placebo: 73 (44.2)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 166 | 165
weeks | 8.3 [8.00 to 9.14] | 12.1 [8.14 to 15.71]
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0100, Log Rank

11. Other Pre Specified Outcome: Durable Remission Week 16 Through Week 52
Description: Remission in a subject from week 16 through week 52.
Time Frame: Week 16 through week 52
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 166 | 165
Participants | 31 | 14
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0077, Cochran-Mantel-Haenszel; Stratified according to anti-TNF agent use (Y/N)

12. Other Pre Specified Outcome: Response at Week 16
Description: as for outcome 2
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 166 | 165
Participants | 79 | 60
Statistical Analysis 1: Comparison: RHB-104 vs Placebo; Test type: Superiority; p = 0.0422, Cochran-Mantel-Haenszel; Stratified according to anti-TNF agent use (Y/N)

13. Other Pre Specified Outcome: Cardiac Safety
Description: Change-from-baseline to week 26 in QTcF (based on cardiac safety report)
Time Frame: Week 26
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 95 | 104
ms | 27.8 [25.91 to 29.74] | 0.2 [-1.67 to 2.06]

14. Other Pre Specified Outcome: Cardiac Safety
Description: Placebo-corrected change-from-baseline to week 52 in QTcF (based on cardiac safety report)
Time Frame: Baseline through week 52
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | RHB-104 | Placebo
Number analyzed (Participants) | 63 | 54
ms | 29.8 [27.57 to 32.02] | -0.8 [-3.16 to 1.57]

ADVERSE EVENTS:
Time Frame: Baseline through 30 days after last dose of study drug, or up to 13 months
Arm/Group | RHB-104 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/165
Serious Adverse Events (participants affected / at risk) | 31/166 | 31/165
Other Adverse Events (participants affected / at risk) | 115/166 | 90/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RHB-104 (N=166) | Placebo (N=165)
Cardiac disorders (Cardiac disorders) | 2 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 19 | 17
General disorders and administration site conditions (General disorders) | 1 | 0
Hepatobiliary disorders (Hepatobiliary disorders) | 2 | 0
Infections and infestations (Infections and infestations) | 4 | 10
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 | 1
Investigations (Investigations) | 2 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal and urinary disorders (Renal and urinary disorders) | 1 | 2
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vascular disorders (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RHB-104 (N=166) | Placebo (N=165)
Crohn's Disease (Gastrointestinal disorders) | 21 | 25
Abdominal Pain (Gastrointestinal disorders) | 24 | 19
Nausea (Gastrointestinal disorders) | 22 | 12
Diarrheoa (Gastrointestinal disorders) | 11 | 8
Vomiting (Gastrointestinal disorders) | 12 | 7
Abdominal tenderness (Gastrointestinal disorders) | 4 | 9
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 9
Influenza (Infections and infestations) | 6 | 10
Viral Upper Respiratory Infections (Infections and infestations) | 7 | 9
Clostridium difficile Infection (Infections and infestations) | 3 | 12
Chromaturia (Renal and urinary disorders) | 42 | 2
Headache (Nervous system disorders) | 16 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 7
Anemia (Blood and lymphatic system disorders) | 10 | 6
Pyrexia (Gastrointestinal disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT01951326/SAP_000.pdf
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT01951326/Prot_001.pdf